CLINICAL TRIAL: NCT07165483
Title: Do Increasing Preoperative Timing of Single Dexmedetomidine Dose Have an Effect on Stress Response of Laryngoscopy and Intubation? A Randomized Controlled Trial
Brief Title: Do Increasing Preoperative Timing of Single Dexmedetomidine Dose Have an Effect on Stress Response of Laryngoscopy and Intubation?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1334/8/25
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Time; Dexmedetomidine; Stress Response; Laryngoscopy; Intubation
MeSH Terms: conditions — Fractures, Stress | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group D20 (Experimental): Patients will receive 0.5µg/kg dexmedetomidine (over 10 min) 20 min before induction of anesthesia then saline (over 10 min) 10 min before induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Group D10 (Experimental): Patients will receive saline (over 10 min) 20 min before induction of anesthesia then 0.5µg/kg dexmedetomidine (over 10 min) 10 min before induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Group C (Placebo Comparator): Patients will receive saline before induction of anesthesia as a control group.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive 0.5µg/kg dexmedetomidine (over 10 min) 20 min before induction of anesthesia then saline (over 10 min) 10 min before induction of anesthesia.
  Arms: Group D20
Drug: Dexmedetomidine — Patients will receive saline (over 10 min) 20 min before induction of anesthesia then 0.5µg/kg dexmedetomidine (over 10 min) 10 min before induction of anesthesia.
  Arms: Group D10
Drug: Saline — Patients will receive saline before induction of anesthesia as a control group.
  Arms: Group C

SUMMARY:
This study aims to evaluate the effect of increasing preoperative timing of single dexmedetomidine on the stress response of laryngoscopy and intubation.

DETAILED DESCRIPTION:
Maintaining hemodynamic stability during surgery is one of the most important tasks because good anesthesia increases the success rate of surgery and improves postoperative prognosis.

Dexmedetomidine, a potent α2-adrenoreceptor agonist, produces not only a sedative-hypnotic effect, but in situations involving cardiac risk, it also produces analgesic effects and an autonomic blocking effect, by acting on a single type of receptor.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.

Exclusion Criteria:

* Severe cardiovascular problems.
* Respiratory disorders.
* Diabetes.
* Hypertension.
* Obesity.
* Allergic reaction to study drugs.
* Patients on antihypertensive medication (α-methyldopa, clonidine, or other α2-adrenergic agonists)
* Medications that affect heart rate (HR) or blood pressure (BP).
* Pregnant.
* Currently breast-feeding women.
* History of sleep apnea.
* Those for emergency procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure | Till the end of the surgery (Up to 2 hours)
  Mean arterial pressure will be recorded at baseline, before induction, after induction, before intubation, after intubation, at 5 minutes, 10 minutes, 15 minutes, and then every 15 minutes until the end of surgery.

SECONDARY OUTCOMES:
Heart rate | Till the end of the surgery (Up to 2 hours)
  Heart rate will be recorded at baseline, before induction, after induction, before intubation, after intubation, at 5 minutes, 10 minutes, 15 minutes, and then every 15 minutes until the end of surgery.
Need for intraoperative fentanyl | Intraoperatively
  Need for intraoperative fentanyl will be recorded.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.